CLINICAL TRIAL: NCT03631849
Title: Epstein-Barr Virus Implication in Peri-implantitis: Towards an Innovative Etiopathogenic Model Involved in Implant-supported Prostheses Loss.
Brief Title: Epstein-Barr Virus Implication in Peri-implantitis: Towards an Innovative Etiopathogenic Model.
Acronym: PERIVIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-AOI-10
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-11

CONDITIONS: Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with peri-implantitis (Experimental)
  Interventions: Procedure: peri implantitis sanitation surgery
- Patients without peri-implantitis (Active Comparator)
  Interventions: Other: Care

INTERVENTIONS:
Procedure: peri implantitis sanitation surgery — an intrasulcular vestibular and lingual / palatal incision with respect to the implant-supported restoration involved is performed, it extends to at least one tooth on either side in order to give laxity to the flap. The use of an incision of discharge will be necessary if the muco-periosteal detachment of the flap (that is to say of full thickness) is considered insufficient to access and unclamp the peri-implant lesion.
  Then, the debridement will be carried out using manual curettes in titanium: the products (waste) removed with this curette will constitute the peri-implant pocket specimens. This sample will be deposited in a Roswell Park Memorial Institute Medium (RPMI) supplemented with serum.The surface of the titanium implant will then be disinfected with betadine, or with hydrogen peroxide for patients with an allergy to polyvidone iodine.
  The flap will then be repositioned and sutured with simple stitches made with a resorbable suture of Vicryl type 5.0.
  Arms: Patients with peri-implantitis
Other: Care — descaling and maintenance of implants
  Arms: Patients without peri-implantitis

SUMMARY:
Peri-implantitis is a high prevalence disease that affects Dental Implants, and can lead to the implant loss if untreated. This condition isn't really well known, and treatments can't provide predictable results. The aim of this study will be to establish a link between the Epstein Barr Virus and the Peri-implantitis, as suggested by recent studies.

DETAILED DESCRIPTION:
Just like the tissues surrounding a natural tooth, the structures around a dental implant, the support of an artificial tooth, can host a severe inflammation, called peri-implantitis. Once it has developed, peri-implantitis is irreversible, and causes the loss of the mucosa and osseous support of the implant, leading inevitably to its loss. The mean prevalence of peri-implantitis is about 10% of all implants, and this pathology affects up to 20% of patients, from 5 to 10 years after surgery. This disease is, therefore, a real public health issue, and a major medico-economic challenge for present-day dentistry. If, like periodontitis (infection/inflammation of the tissues surrounding a natural tooth), peri-implantitis seems to be multifactorial, it is proven that a diverse and pathogenic bacterial flora colonizes the peri-implant tissues and plays a major role in bone loss. Poor oral hygiene and uncontrolled diabetes are among the known risk factors. Furthermore, a link has been clearly established between an antecedent of periodontitis and the risk of contracting peri-implantitis. However, this infection tends to progress slowly, before any clinical symptoms appear (e.g. suppuration, pain, implant mobility) which means that the pathology is advanced and is, most often, going to lead to implant loss. At present only very early diagnosis and treatment (at the mucositis stage) are able to stabilize the evolution of this disease. Moreover, present-day treatments (surgical debridement, with or without bone regeneration) are not easily reproducible, leading to an unfavorable prognosis. If prevention of peri-implant disease (follow-up examination, radiography, peri-implant probing and perfect oral hygiene) is essential to maintaining healthy peri-implant tissues, it does not guarantee the implant's sustainability. Indeed, peri-implant tissues are scar tissues, less well vascularized than periodontal tissues, and without the periodontal ligament, which links the tooth to the surrounding bone and plays an immune-protective role. Thus, peri-implant sites are less well-organized to resist oral bacterial assault, which certainly explains the high prevalence of peri-implant diseases. No correlation was found between the implant surface treatment or the implant design, and the development of a peri-implantitis.

However, neither the onset, nor the trigger, nor even the mechanisms underlying the progression of peri-implantitis are clearly understood at the moment. Even if the inflammatory role of bacterial dysbiosis remains predominant, several lines of evidence suggest that the bacterial etiology is not sufficient to totally explain the pathology, especially the initial stages, its non-reversible inflammatory nature, and the failure of antibiotic therapies.

A possible synergy between the peri-implant bacteria pathogenicity and the replication/activation of endogenous herpes virus seems to be a hypothesis in the development of peri-implantitis. This model of viro-bacterial synergy represents one of the major mechanistic advances concerning periodontitis.

A previous study, (Vincent et al., 20135), in particular, proved that the Epstein-Barr Virus (EBV) infection, an ubiquitous human herpesvirus with chronic oral replication, was detectable in healthy gums, and grew significantly in the deepest periodontal pockets. Moreover, this study clearly established for the first time that the epithelial cells surrounding periodontally affected teeth were frequently infected by EBV, and showed a high susceptibility to apoptosis. This epithelial damage characterized by the death of infected cells, certainly contributes to the loss of attachment between bone and teeth, promoting bacterial invasion and serious inflammation.

There is still little data on the involvement of EBV in peri-implantitis, but it has been recently proved that the virus is present twelve times more often in an affected peri-implant area than in a healthy area, with a positive predictive value between EBV and peri-implantitis of 90%. Moreover, EBV has been associated to the most severe cases of peri-implantitis. In addition, a significant correlation between EBV and mucositis (reversible initial stage of peri-implant inflammation) seems to exist. If it is accepted that untreated mucositis systematically evolves into irreversible periimplantitis any early identification of mucositis markers would allow treatment at an early stage of the disease. Finally, this data is also supported by our own recent preliminary results that show the presence of EBV in peri-implantitis sites.

All these results point to the proposition that EBV may play a role in the onset and/or the development of peri-implantitis. The objective of this research project is to test this hypothesis and see if the results for periodontitis could be applied to peri-implantitis.

This is an original project that it now seems essential to investigate as part of a clinical study. It draws on the already established expertise of the research laboratory of the Faculty of Dentistry (MICORALIS, directed by Dr Alain Doglio), associated with Nice University Hospital Dental Department, and is the continuity of Dr Vincent's work. The evidence of an implication of EBV in peri-implantitis could open a way to identifying a new early pathogenic marker and lead to a new antiviral therapeutic approach, which could, in time, prevent implant loss.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Patient with at least one dental implant with a fixed implant-supported prostheses
* Patient with a peri-implantitis
* (Patient with healthy dental implant for control group)
* patients having read and understood the information note on the study and signed the informed consent form.
* patients affiliated to the social security system.

Exclusion Criteria:

* Patient with severe hematologic disease
* Patients with previous or current acute illness or severe chronic cardiovascular, renal, hepatic, gastrointestinal, allergic, endocrine, neuro-psychiatric, considered by the investigator to be incompatible with the conduct of the study.
* Patients treated with retinoids, oral bisphosphonates, oral anticoagulants or anticonvulsants.
* Patient have or have had cancer of the upper aerodigestive tract treated by radiotherapy.
* Patient taking a steroidal or non-steroidal anti-inflammatory, anti-cancer or immunosuppressive chemotherapy in the last 6 months.
* Patient monitoring considered difficult by the investigator.
* Patient with oral dermatitis or adverse occlusion.
* Patient with autoimmune disease
* Patient with a linguistic or mental incapacity to understand information
* Patient trust under curators or judicial protection
* Patient participating in another clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2025-10-28 (Actual); Study Completion 2025-10-28 (Actual)

PRIMARY OUTCOMES:
Correlate the Epstein-Barr Virus (EBV) levels of peri-implant sites with the presence of peri-implantitis | At inclusion, at surgery and 1, 6, 12 and 18 months post-surgery
  The Epstein-Barr Virus (EBV) levels in periodontal sample is measured through quantitative Polymerase Chain Reaction (PCR) of their viral genomes, throughout patient follow-up.

SECONDARY OUTCOMES:
Correlate cellular viral load to depth of peri-implant pocket | At inclusion, at surgery and 1, 6, 12 and 18 months post-surgery
  The cellular viral load is the percentage of epithelial cells infected with Epstein-Barr Virus (EBV) and will assessed by in situ hybridation in peri-implant pocket samples. It will be correlated to the depth of peri-implant pocket.
Correlate cellular viral load to peri-implantite treatment failure (recurrence) | At 1, 6, 12 and 18 months post-surgery
  Recurrence will be defined by the presence of additional radiographic bone loss (compared to the last visit), increased of peri-implant pocket depth (in millimeters) and the présence of bleeding or suppuration. Cellular viral load is defined at the first secondary outcome measure.
Correlate cellular viral load to local inflammatory response during follow-up | At inclusion, at surgery and 1, 6, 12 and 18 months post-surgery
  The local inflammatory response will be assessed by the quantification of inflammatory cytokines in peri-implant pocket cells. The quantification will be done with the enzyme-linked immunosorbent assay (ELISA). Cellular viral load is defined at the first secondary outcome measure.
Correlate cellular viral load to the presence of virulent bacteria | At 1, 6, 12 and 18 months post-surgery
  Virulent bacteria will be assessed by quantitative Polymerase Chain Reaction (PCR) of their viral genomes on bacterial plaque sample
Characterize Epstein-Barr Virus (EBV)-infected cell types | At 1, 6, 12 and 18 months post-surgery
  Epstein-Barr Virus (EBV)-infected cell types will be caracterized using fluorescent co-immunomarkings on peri-implant pocket samples and gum cuts.
Study the virological profile of the expression of viral proteins EBV in lesional site | At 1, 6, 12 and 18 months post-surgery
  The virological profile of the expression of viral proteins EBV in lesional site will be assessed using immunofluorescence and reverse transcription associated to quantitative Polymerase Chain Reaction (RT-qPCR).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France, France